CLINICAL TRIAL: NCT04914598
Title: A Randomized, Controlled, Double-blind, Multi-center Phase Ⅲ Registration Clinical Study of Combined Cisplatin Versus Placebo Combined With Intracavitary Cisplatin Injection in the Treatment of Malignant Pleural Effusions
Brief Title: A Phase Ⅲ Clinical Study of Combined Cisplatin Versus Placebo Combined With Intracavitary Cisplatin Injection in the Treatment of Malignant Pleural Effusions
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-372-ENDO-301
Record Dates: First submitted 2021-05-27; First posted 2021-06-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENDOSTAR combined with cisplatin (Active Comparator)
  Interventions: Drug: ENDOSTAR，cisplatin
- Placebo combined with cisplatin (Placebo Comparator)
  Interventions: Drug: Placebo , cisplatin

INTERVENTIONS:
Drug: ENDOSTAR，cisplatin — After sufficient puncture and drainage or drainage, use Endo® (45mg/time in thoracic cavity, 60mg/time in abdominal cavity) + cisplatin (40mg/time) intracavitary injection, administration on 1, 4, and 7 days, 3 times as a course of treatment
  Arms: ENDOSTAR combined with cisplatin
Drug: Placebo , cisplatin — Placebo , cisplatin
  Arms: Placebo combined with cisplatin

SUMMARY:
Malignant Pleural Effusion or Ascites is a common complication of malignant tumor, The objective of this study is to compare the efficacy of Endostar/cisplatin with placebo/cisplatin in patients with malignant pleural effusion or ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed cancer of any primary tumor type, Patients with Malignant Pleural Effusion or Ascites who remain poorly controlled after at least one systemic antitumor therapy and at least one local therapy (intracavitary administration of chemotherapeutic agents and/or biological response modulators, other than cisplatin.)
2. At least a medium amount of malignant pleural effusion or ascites conformed by confirmed by B ultrasound, Clinical judgment requires local therapy.
3. Karnofsky Performance Status ≥60
4. Life expectancy of at least 3 months
5. Adequate hematologic, cardiac, renal, and hepatic function
6. The serum pregnancy test of female subjects of childbearing age during the screening period was negative; With a fertile female/male subjects must be willing to throughout the study period (i.e., for the first time since the drug delivery to the end of the study drug dosing after 90 days) to take reliable contraceptive methods, including but not limited to: abstinence, male partners have accepted vasectomy, female sterilization, intrauterine device effectively and effective birth control pills.

Exclusion Criteria:

1. Participating in or receiving investigational treatment in another clinical trial within 4 weeks prior to first dosing, or participating in a device clinical trial within 4 weeks Evidence of bleeding diathesis, serious infection
2. Received systemic antitumor therapy or intraperitoneal drug therapy within 14 days of the first intracavitary administration;
3. Endostatin, bevacizumab, Ramucirumab, and other antiangiogenic agents or cisplatin were used for local therapy
4. Has not recovered from any adverse event due to any intervention to ≤1 prior to initial administration (except for hair loss, hearing loss, and neurological or endocrine disorders of ≤2 requiring alternative treatment)
5. Had undergone medium to major surgery other than diagnosis or biopsy within 28 days prior to first administration, or who were expected to undergo major surgery during the study period
6. Bilateral pleural effusion or enveloped pleural effusion or ascite
7. With severe COPD or a history of intestinal adhesions
8. uncontrolled primary brain tumor or central nerve metastatic tumor with significant intracranial hypertension or neuropsychiatric symptoms
9. Active infections that require systemic treatment
10. Pregnant or lactating women
11. history of illness, treatment, or laboratory abnormality that may interfere with the outcome of the study and prevent subjects from participating fully in the study, or participation is not considered by the investigator to be in the subjects' best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Puncture/drainage-Free Survival, PuFS | From the date of the end of experiment therapy to the next Puncture /drainage or death from any cause, up to 6 months
  Compared with placebo combined with intracavitary cisplatin injection, use Puncture/drainage-Free Survival (Puncture/drainage-Free Survival, PuFS) as an indicator to evaluate Endo® combined with cisplatin intracavitary injection in the treatment of malignant pleural or ascites effusion Efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, Doctor, Study Chair — Shanghai East Hospital of Tongji University; Jin Li, Doctor, Study Chair — Shanghai East Hospital of Tongji University
Locations (1):
- Yan Xie, Nanjing, China

IPD SHARING:
Plan to Share IPD: No